CLINICAL TRIAL: NCT00008086
Title: A Phase I Trial of Subcutaneous And/Or Oral Calcitriol [(1,25-COH)2D3] and Carboplatin in Advanced Solid Tumors
Brief Title: Calcitriol Plus Carboplatin in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura A. Pollice, Clinical Research Manager, University of Pittsburgh
Purpose: Treatment
Other Study IDs: 97-004; CDR0000068374 (Registry Identifier: PDQ (Physician Data Query)); PCI-IRB-970532; NCI-G00-1885
Record Dates: First submitted 2001-01-06; First posted 2003-09-04 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Brain and Central Nervous System Tumors; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent adult brain tumor; adult brain stem glioma; adult craniopharyngioma; adult medulloblastoma; adult meningioma; adult glioblastoma; unspecified adult solid tumor, protocol specific; adult anaplastic astrocytoma; adult myxopapillary ependymoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult central nervous system germ cell tumor; adult pilocytic astrocytoma; adult subependymoma; adult ependymoblastoma; adult pineocytoma; adult pineoblastoma; adult meningeal hemangiopericytoma; adult choroid plexus tumor; adult grade III meningioma; adult oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Craniopharyngioma; Medulloblastoma; Meningioma; Glioblastoma; Astrocytoma; Ependymoma; Oligodendroglioma; Glioma; Glioma, Subependymal; Neuroectodermal Tumors, Primitive; Pinealoma; Choroid Plexus Neoplasms; Gliosarcoma | interventions — Calcitriol; Carboplatin

INTERVENTIONS:
Dietary Supplement: calcitriol
Drug: carboplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Calcitriol may help solid tumor cells develop into normal cells. Combining calcitriol with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of calcitriol combined with carboplatin in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated doses of calcitriol and carboplatin, when given in combination, in patients with advanced solid tumors.
* Determine the toxic effects of this regimen in these patients.
* Determine the effect of calcitriol on the pharmacokinetics of carboplatin in these patients.
* Correlate the pharmacokinetics of carboplatin with the myelosuppression following this regimen in these patients.
* Determine the safety and efficacy of this regimen in patients with malignant glioma.

OUTLINE: This is a dose-escalation study. Patients are stratified according to disease (brain tumor vs other solid tumor) and accrued in parallel. Patients are assigned to one of two treatment groups.

* Group 1: Patients receive carboplatin IV over 20-30 minutes on day 1 and calcitriol subcutaneously (SC) or orally daily on days 2-4 for the first course only. For subsequent courses, patients receive calcitriol SC or orally daily on days 1-3 and carboplatin IV over 20-30 minutes on day 3.
* Group 2: Patients receive calcitriol SC or orally daily on days 1-3 and carboplatin IV over 20-30 minutes on day 3 for the first, third, and subsequent courses. For the second course only, patients receive carboplatin IV over 20-30 minutes on day 1 and calcitriol SC or orally daily on days 2-4.

In both groups, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Sequential dose escalation of calcitriol is followed by sequential dose escalation of carboplatin. Cohorts of 3-6 patients receive escalating doses of calcitriol and then carboplatin until the maximum tolerated dose (MTD) of the combination is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 18-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumor that is not curable by standard therapy, including glioma and other brain tumors
* Brain metastases allowed following definitive radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 4 times normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min
* Creatinine no greater than 2.0 mg/dL
* Calcium no greater than 10.5 mg/dL

Cardiovascular:

* No unstable angina
* No symptomatic coronary artery disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of barrier contraception AND 1 form of hormonal contraception for at least 1 week before, during, and for at least 2 weeks after study
* No active infection
* No other concurrent serious condition

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy (regional or systemic)

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* No concurrent glucocorticoids as antiemetics
* Concurrent exogenous glucocorticoids allowed for treatment of gliomas or other brain tumors

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* Dietary calcium intake of no more than 200-250 mg/day beginning 48 hours before each course and continuing for 7 days
* No concurrent dairy products, green leafy vegetables, molasses, baking powder, fortified cereals, and dry peas and beans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-01; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh K. Ramanathan, MD, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States